CLINICAL TRIAL: NCT00408291
Title: Evaluation of the Winsta PH Osteosynthesis Device in the Treatment of Three- and Four-Part Fractures of the Proximal Humerus A Prospective Migration and Bone Density Study
Brief Title: Evaluation of Treatment of Fractures of the Humerus With a Plate.
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 20060166
Record Dates: First submitted 2006-12-05; First posted 2006-12-06 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Fracture
Keywords: fracture; shoulder; bone density; healing
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Winsta PH osteosynthesis device (Fischer Medical)for treatment of humeral fracture
  Interventions: Procedure: Winsta PH osteosynthesis device

INTERVENTIONS:
Procedure: Winsta PH osteosynthesis device — The Winsta PH osteosynthesis device have been developed for use in treatment of proximal humerus fractures.
  Other Names: Winsta PH osteosynthesis device (Fischer Medical)

SUMMARY:
The purpose of this study is to study with the use of clinical and radiological parameters the treatment of three-part and four-part fractures with the Winsta PH osteosynthesis device (Fischer Medical).

DETAILED DESCRIPTION:
We shall measure the following clinical parameters with the help of the Constant Shoulder Score (CSS) and Western Ontario Osteoarthritis of the Shoulder Index (WOOS):

1. Pain
2. Activities of Daily Living (ADL)
3. Range of Motion (ROM)
4. Muscle strength

We shall measure the following radiologic parameters:

1. Healing (migration) of tuberculum majus and minus measured with use of MB-RSA
2. Plate migration with use of MB-RSA
3. Bone density in the proximal humerus measured with Dual Energy X-ray Absorptiometry (DEXA)
4. Correlation between bone density and prosthesis migration (and tuberculum migration)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with three-part and four-part proximal humeral fractures
2. Aged 50 years or older and fit
3. Informed, written consent
4. A functioning shoulder preoperatively -

Exclusion Criteria:

1. Patients found unsuitable preoperatively for a shoulder Philos Plate
2. Patients aged 85 or older
3. Patients with rheumatoid arthritis
4. Patients who previously had undergone shoulder plastic or other major shoulder surgery
5. Patients unable to avoid NSAID after surgery
6. Patients requiring regular systemic steroid treatment
7. Female patients taking hormone substitution
8. Female patients in the fertile age range who do not use safe anti-conception (oral contraception, intrauterine devices, depot gestagens, vaginal hormone rings)
9. Patients with metabolic bone disease -

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be included at 2 orthopaedic departments at 2 hospitals
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
Healing (migration) of tuberculum majus and minus measured with use of Model-Based Roentgen Stereophotogrammetric Analysis (MB-RSA) | five years
  Migration of the tubercles measured with Model-Based Roentgen Stereophotogrammetric Analysis (MB-RSA)

SECONDARY OUTCOMES:
Correlation between bone density and prosthesis migration (and tuberculum migration) | five years
Range of Motion (ROM) | five years
Muscle strength | five years
Activities of Daily Living (ADL) | five years
Bone density in the proximal humerus measured with Dual Energy X-ray Absorptiometry (DEXA) | five years

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Soballe, Professor, Study Director — Orthopaedic Department, Aarhus University Hospital
Locations (1):
- Orthopaedic Department K, Silkeborg Hospital, Silkeborg, Denmark

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196